CLINICAL TRIAL: NCT03551314
Title: Effects of Two Modalities of Non-invasive Ventilation on Breathing Pattern Variables of Preterm Neonates of Very Low Weight After Extubation
Brief Title: Effects of Two Modalities of Non-invasive Ventilation After Extubation in Very Low Birth Weight Neonates
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Minas Gerais (Other)
Collaborators: Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government)
Responsible Party: Principal Investigator, Veronica Franco Parreira, Full Professor, Federal University of Minas Gerais
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CAAE: 67787917.7.0000.5149
Record Dates: First submitted 2018-05-15; First posted 2018-06-11 (Actual); Last update posted 2019-02-21 (Actual); Status verified 2019-02

CONDITIONS: Preterm Infant
Keywords: Non-invasive ventilation; Preterm infant; Breathing pattern
MeSH Terms: conditions — Premature Birth | interventions — Continuous Positive Airway Pressure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nasal Intermittent Positive Pressure (Active Comparator): In this group, soon after extubation, the newborns will be studied initially in NIPPV for one hour. Infants will be studied in supine while in their incubator.
  NIPPV: Nasal Intermittent Positive Pressure Ventilation
  Interventions: Other: Nasal Intermittent Positive Pressure
- Continuous Positive Airway Pressure (Active Comparator): In this group, soon after extubation, the newborns will be studied initially in CPAP for one hour. Infants will be studied in supine while in their incubator.
  CPAP: Continuous Positive Airway Pressure
  Interventions: Other: Continuous Positive Airway Pressure

INTERVENTIONS:
Other: Nasal Intermittent Positive Pressure — - NIPPV The following parameters: inspiratory pressure = 15 cmH2O / final expiratory positive pressure = 6 cmH2O / inspiratory time = 0.40 / flow = 6-8 L.min-1 / respiratory rate = 24.
  Respiratory inductive plethysmography is used to evaluate breathing pattern (tidal volume, respiratory rate, minute ventilation, mean inspiratory flow) and chest wall motion (labor breathing index - LBI, phase relation in inspiratory breathing - PhRIB, phase relation in expiratory breathing - PhREB, total phase relation - PhRTB and phase angle).
  Arms: Nasal Intermittent Positive Pressure
Other: Continuous Positive Airway Pressure — - CPAP The following parameters: pressure of 6 cmH2O, with flow of 6-8L/min.
  Respiratory inductive plethysmography is used to evaluate breathing pattern (tidal volume, respiratory rate, minute ventilation, mean inspiratory flow) and chest wall motion (labor breathing index - LBI, phase relation in inspiratory breathing - PhRIB, phase relation in expiratory breathing - PhREB, total phase relation - PhRTB and phase angle).
  Arms: Continuous Positive Airway Pressure

SUMMARY:
The objective of this study is to evaluate the effects of continuous positive airway pressure and nasal intermittent positive pressure ventilation on breathing pattern variables of very low birth weight neonates immediately after extubation.

DETAILED DESCRIPTION:
The effects of non-invasive ventilation on the respiratory function of neonates have not been fully elucidated. Currently, two modalities of non invasive ventilation are commonly used in Brazilian neonatal intensive care units: continuous positive airway pressure (CPAP) and nasal intermittent positive pressure ventilation (NIPPV). In this study, it was hypothesized that NIPPV will improve tidal volume when compared to CPAP. The objective of this study is to evaluate the effects of continuous positive airway pressure and nasal intermittent positive pressure ventilation on breathing pattern variables of very low birth weight neonates immediately after extubation. Soon after extubation, the neonates will be randomized into the CPAP-NIPPV (sequence 1) or the NIPPV-CPAP (sequence 2). The sequence will be assigned at random using sealed envelopes. Respiratory inductive plethysmography will be used to evaluate the breathing pattern (tidal volume, respiratory rate, minute ventilation, mean inspiratory flow) and chest wall motion (labor breathing index, inspiratory phase relation, expiratory phase relation, total phase relation and phase angle). Student t tests for paired samples will be used and the Wilcoxon test according to the data distribution. A significance level of 5% will be adopted. The analyzes will be performed by StatisticalPackage software for the Social Sciences® (SPSS, Chicago, IL, USA), version 17.0 for Windows.

ELIGIBILITY:
Inclusion Criteria:

* Presented gestational age less than or equal to 32 weeks and weight less than or equal to 1,500 g;
* Stability from an hemodynamic point of view (without use of amines);
* Have undergone invasive mechanical ventilation;
* Absence of congenital heart diseases and / or other congenital anomalies (myelomeningocele, gastroschisis and / or omphalocele) or chromosomal abnormalities;
* Absence of any condition that requires surgery in the neonatal period.

Exclusion Criteria:

* Presented air leak syndrome (pneumothorax, pneumomediastinum); upper airway obstruction after extubation and non-scheduled extubation.

Max Age: 32 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 17 (Actual)
Dates: Start 2017-05-26 (Actual); Primary Completion 2018-07-26 (Actual); Study Completion 2018-07-26 (Actual)

PRIMARY OUTCOMES:
Tidal volume | Measure during the two non-invasive ventilation strategies. Tidal volume will be measured for 2 hours, one hour in continuous positive airway pressure and one hour in nasal intermittent positive pressure ventilation.
  Defined as the volume of air entering or exiting the lungs during each breath - in millilitres.

SECONDARY OUTCOMES:
Respiratory rate | Measure during the two non-invasive ventilation strategies. Respiratory rate will be measured for 2 hours, one hour in continuous positive airway pressure and one hour in nasal intermittent positive pressure ventilation.
  Breaths per minute
Minute ventilation | Measure during the two non-invasive ventilation strategies. Minute ventilation will be measured for 2 hours, one hour in continuous positive airway pressure and one hour in nasal intermittent positive pressure ventilation.
  Computed from tidal volume multiplied by respiratory rate, in liters/minute
Mean inspiratory flow | Measure during the two non-invasive ventilation strategies. Mean inspiratory flow will be measured for 2 hours, one hour in continuous positive airway pressure and one hour in nasal intermittent positive pressure ventilation.
  Is a estimation of respiratory center drive activity. The higher its value, the greater the drive and vice-versa.
Labored Breathing Index (LBI) | Measure during the two non-invasive ventilation strategies. Labor breathing index (LBI) will be measured for 2 hours, one hour in continuous positive airway pressure and one hour in nasal intermittent positive pressure ventilation.
  This is a measure of chest wall coordination. This is the Labored Breathing Index (LBI) of a breath that takes into account phase and amplitude of the ribcage and abdomen traces. It is computed as the ratio of the sum of the integrals of the absolut values of the derivatives of the inspiratory limbs of ribcage and abdomen excursions divided by the corresponding integral of the derivative of the inspiratory limb of the tidal volume deflection. This measure of thoracoabdominal coordination is computed on a breath by breath basis. Perfect thoracoabdominal coordination produces an LBI of 1.0. In babies or adults who are relaxed and awake or in Quiet State, LBI lies between 1.0 and 1.2 but no systematic study of the normal values of LBI as a function of sleep stage and body posture has yet been undertaken. In Active State, thoracoabdominal discoordination generally is associated with elevated LBI values.
Phase relation in inspiratory breathing (PhRIB) | Measure during the two non-invasive ventilation strategies. Phase relation in inspiratory breathing will be measured for 2 hours, one hour in continuous positive airway pressure and one hour in nasal intermittent positive pressure ventilation.
  This express the percentage agreement between direction of ribcage and abdomen movements during the inspiratory phase of breath.
Phase relation in expiratory breathing | Measure during the two non-invasive ventilation strategies. Phase relation in expiratory breathing will be measured for 2 hours, one hour in continuous positive airway pressure and one hour in nasal intermittent positive pressure ventilation.
  This express the percentage agreement between direction of ribcage and abdomen movements during the expiratory phase of breath.
Phase relation in total breathing | Measure during the two non-invasive ventilation strategies. Phase relation in total breathing will be measured for 2 hours, one hour in continuous positive airway pressure and one hour in nasal intermittent positive pressure ventilation.
  This express the percentage agreement between direction of ribcage and abdomen movements during the entire breath cycle.
Phase angle | Measure during the two non-invasive ventilation strategies. Phase angle will be measured for 2 hours, one hour in continuous positive airway pressure and one hour in nasal intermittent positive pressure ventilation.
  The phase angle is computed from Lissajous loops between ribcage and abdomen excursions on a breath by breath basis.

CONTACTS AND LOCATIONS:
Overall Officials: Verônica F Parreira, PhD, Principal Investigator — Federal University of Minas Gerais
Locations (2):
- Brazil (2):
  - Hospital das Clínicas da UFMG, Belo Horizonte, Minas Gerais
  - Laboratório de Avaliação e Pesquisa em Desempenho Cardiorrespiratório da UFMG, Belo Horizonte, Minas Gerais

IPD SHARING:
Plan to Share IPD: No